CLINICAL TRIAL: NCT02858778
Title: A Randomized Allocation of Palliative Care Consultation in the Emergency Department Compared to Usual Practice
Brief Title: Timing of Acute Palliative Care Consultation in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wayne State University (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Robert Zalenski, Principle Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BCBSMF PSACO
Record Dates: First submitted 2016-07-20; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Organ Failure; End Stage Cardiac Failure; End Stage Chronic Obstructive Airways Disease; Chronic Kidney Disease Stage 5; Hepatic Encephalopathy; Sepsis; Dementia; Multiple Sclerosis; Parkinson's Disease; In-Hospital Cardiac Arrest; Solid Organ Cancer
Keywords: Palliative Care; Emergency Department
MeSH Terms: conditions — Multiple Organ Failure; Renal Insufficiency, Chronic; Hepatic Encephalopathy; Sepsis; Dementia; Multiple Sclerosis; Parkinson Disease; Emergencies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Interventional group (Ig) (Experimental): The interventional group (Ig) will have an early palliative care consultation ordered during their stay in the emergency department.
  Interventions: Other: Early order of palliative care consultation
- Control group (Cg) (No Intervention): The control group will be treated as standard of care. Palliative care consultations may or may not be ordered at the attending physician's discretion.

INTERVENTIONS:
Other: Early order of palliative care consultation
  Arms: Interventional group (Ig)

SUMMARY:
A prospective randomized controlled trial studying the ordering of palliative care consultations in the emergency department (Ig) versus later palliative care consultations in the hospital--ICU or hospital ward(Cg). Patients will be randomly allocated to Ig or Cg with a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 65 years old
* Treated in a resuscitation room for unstable vital signs or respiratory compromise
* One or more of the following:
* Advanced or metastatic solid organ cancer
* End stage organ failure of the heart, lung/COPD, kidney on dialysis, hepatic encephalopathy
* Suspected sepsis
* Advanced dementia, end-state multiple sclerosis or Parkinson's disease
* Status post cardiac arrest with coma (Glascow coma score <7)
* Patient is from a skilled nursing facility

Exclusion Criteria:

* Lack decision capacity and have no relative available during ED stay to consent to the study (legally authorized representative-LAR)
* Enrolled in hospice care prior to randomization
* A copy of a completed advance directive which names a designated proxy provided physically to the medical team prior to randomization
* Wearing a DNR bracelet
* Have been previously enrolled in this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The difference in the percentage of patients with a completed advance directive (AD) in Ig vs.Cg | 1 year

SECONDARY OUTCOMES:
The proportion of billed CMS ACP-CPT codes in Ig vs. Cg | 30 days from enrolled patients' hospital discharge
  The proportion of patients who received an ACP CMS billing codes (which took effect in January 2016), in Ig vs. Cg will be evaluated using one or both of the new CPT codes for Advance care planning (ACP) services…including the explanation and discussion of advance directives such as standard forms (with the completion of such forms, when performed) by the physician or other qualified health profession; first 30 (15-45)minutes, face to face with the patients, family member(s) and/or surrogate Code 99497; and each additional 30 (46-75 minutes)-Code 99498 (Federal Register, 2015).
Matches of care received to patient-specific preferences in Ig vs. Cg | 1 year
  The investigators will align treatment preferences with medical orders, replicated as reported in the study by Mack et al. Proportions of patients coded as having a match will be compared across the treatment and control groups. For everyone who gets ACP during the study, patients or their surrogates will be asked by a member of the care team-either palliative care if they are consulted, or the hospital based care team if they are not: "If you could choose, would you prefer (a) treatment that focuses on attempting to extend your time as much as possible, even if doing so means more pain and discomfort, or (b) a plan of care that focuses on relieving pain and discomfort and improving quality of life, even though that may mean not living as long.
Patient/family satisfaction with care in Ig vs. Cg | Baseline
  This outcome will be measured on a continuous scale. The net-promoter score will be measured at baseline (at randomization) and at hospital discharge for a change in value. It is measured on a scale of 1-10. Whoever signs the consent (patient of LAR) will be asked the net promoter score, and that will be reassessed by them at discharge, unless the patient has died-and the variable will then be recorded as missing. The PSQ will be administered by research assistants at the time of the patient's discharge. If the patient is incapacitated, then it will be asked of the patient's closest family caregiver. So PSQ is only at discharge of patient or available, most involved, family caregiver.
Amount of hospice referrals in Ig vs. Cg | 1 year
Hospital total direct costs for the index visit in Ig vs. Cg | 1 year
Hospital and ICU length of stay in Ig vs. Cg | 1 year
Average days in hospice in Ig vs. Cg | 1 year
Hospital margin contribution for the index visit in Ig vs. Cg | 1 year
Time to consultation in Ig vs. Cg groups | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zalenski, M.D., M.A., Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - Detroit Medical Center Detroit Receiving Hospital, Detroit, Michigan
  - Detroit Medical Center Sinai Grace Hospital, Detroit, Michigan